CLINICAL TRIAL: NCT02635789
Title: A Double-blind, Randomized, Placebo-controlled Phase III Trial to Investigate the Efficacy and Safety of NPC-12G Gel (Topical Formulation of Sirolimus) to Angiofibroma and Other Skin Lesions in Patients With Tuberous Sclerosis Complex
Brief Title: Phase III Trial of Topical Formulation of Sirolimus to Skin Lesions in Patients With Tuberous Sclerosis Complex (TSC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nobelpharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NPC-12G-1
Record Dates: First submitted 2015-12-15; First posted 2015-12-21 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Tuberous Sclerosis; Angiofibroma; Hypomelanotic Macule; Plaque
Keywords: Sirolimus; Skin lesions; TSC; Tuberous Sclerosis Complex; NPC-12G; Angiofibroma; Hypomelanotic macule; Plaque
MeSH Terms: conditions — Tuberous Sclerosis; Angiofibroma; Plaque, Amyloid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NPC-12G gel (Experimental): NPC-12G gel is containing 0.2% Sirolimus
  Interventions: Drug: NPC-12G gel
- Placebo gel (Placebo Comparator): Placebo gel is matched ingredient with NPC-12G gel
  Interventions: Drug: Placebo gel

INTERVENTIONS:
Drug: NPC-12G gel — NPC-12G gel is administered topically twice a day for 12 weeks
  Arms: NPC-12G gel
Drug: Placebo gel — NPC-12G gel placebo is administered topically twice a day for 12 weeks
  Arms: Placebo gel

SUMMARY:
The purpose of this trial is to evaluate the efficacy and safety of NPC-12G gel (topical formulation of sirolimus) versus placebo gel to facial angiofibroma and other skin lesions in patients with tuberous sclerosis complex (TSC)

DETAILED DESCRIPTION:
Tuberous Sclerosis Complex (TSC) is an autosomal dominant hereditary disease that causes benign tumors on the almost whole body (including skin, brain, kidney, lung and heart), behavior disorder as autism, mental retardation and neurologic symptom as epilepsy. Angiofibroma is TSC-specific facial skin lesions, and hamartoma caused by increase of the component of skin connective tissues and blood vessels. Other skin lesions due to TSC are white macule(hypomelanotic macule), plaque, shagreen patch and ungual fibromas. Current therapeutic methods for angiofibroma are laser or surgical treatments, but there are problems as many relapses, deficiency of evidence, change of pigment, scar and risk of infection.

This will be a multicenter, double-blind, randomized, placebo-controlled parallel group trial. The trial has three phases; the screening phase, double-blinded treatment phase, and post-treatment phase. The screening phase comprises a screening visit where subject's initial eligibility will be evaluated. During double-blinded treatment phase, patients who meet all entry criteria for the trial will be randomized into two groups, and they will apply 0.2% NPC-12G gel or placebo gel topically twice a day for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 3 years old or greater at the time of informed consent
2. Patients who are diagnosed as definite diagnosis according to diagnostic criteria for tuberous sclerosis complex (International Tuberous Sclerosis Complex Consensus Conference 2012)
3. Patients with three or more papules of angiofibroma ( >= 2 mm in diameter with redness in each) on the face at screening tests
4. Patients who are not suitable for therapy with laser or surgery, or who do not want therapy with laser or surgery
5. Patients or his/her guardian who give a written informed consent in understanding and willingness after having received enough explanation of the test drug and the current trial plan

Exclusion Criteria:

1. Patients who are hard to apply the test drug topically with keeping compliance
2. Patients with clinical findings such as erosion, ulcer and eruption on or around the lesion of angiofibroma, which may affect assessment of safety or efficacy
3. Patients who are hard to be taken pictures of their lesions adequately in such cases that they may not follow instruction of stillness
4. Patients with a history of hypersensitivity to alcohol or allergy to sirolimus
5. Patients who have complications such as malignant tumor, infection, serious heart disease, hepatic function disorder, renal function disorder or blood disorders which severity are considered by investigator as grade 2 or more severe with reference to ''Concerning classification criteria for seriousness of adverse drug reactions of medical agents''
6. Patients who have complications such as diseases unsuitable for the trial participation, for examples, uncontrolled diabetes (fasting blood glucose level >140 mg/dL or postprandial blood glucose level > 200 mg/dL), dyslipidemia (cholesterol level > 300 mg/dL or > 7.75 mmol/L, triglycerides level > 300 mg/dL or > 3.42 mmol/L), etc.
7. Patients who have taken drugs with mTOR inhibitory action including sirolimus, everolimus or temsirolimus within 12 months before the initial registration
8. Patients who have applied topical tacrolimus on the lesion of angiofibroma within 3 months before the initial registration
9. Patients who have received therapy with laser or surgery to the lesion of angiofibroma within 6 months before the initial registration
10. Female patients who may be pregnancy or are lactating
11. Patients who cannot agree to take appropriate measures of contraception until completion of post-treatment phase or follow-up period after discontinuation from informed consent
12. Patients who have participated in other clinical trial and have taken a trial drug within 6 months before the initial registration
13. Others, patients who are considered by the investigator as unsuitable for participation in the trial

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Improvements in angiofibroma | 12 weeks
  Improvements comparing with baseline is assessed using photograph by the central photo-judgement committee

SECONDARY OUTCOMES:
Improvements in angiofibroma | Week 4 and 8 and follow-up Week 16
  Improvements comparing with baseline is assessed using photograph by the central photo-judgement committee
Improvements in angiofibroma | Week 4, 8, 12 and follow-up Week 16
  Improvements comparing with baseline is assessed by the investigator
Improvements in redness of angiofibroma | Week 4, 8, 12 and follow-up Week 16
  Improvement comparing with baseline is assessed by the central photo-judgement committee and the investigator
Improvements in hypomelanotic macule and plaque of upper neck | Week 4, 8, 12 and follow-up Week 16
  Improvement comparing with baseline is assessed by the central photo-judgement committee and the investigator
The rate of patients who are evaluated as ''improvement'' or more (improvement rate) in primary outcome measure and in secondary outcome measures above outcome 1 to 5 | Week 4, 8, 12 and follow-up Week 16
Change in total score from baseline for DLQI and CDLQI | Week 4, 8, 12 and follow-up Week 16
  DLQI for subjects 16 years old and greater, or CDLQI for children of less than 16 years old is assessed by patients
Adverse events | 16 weeks
  Adverse events during the study period
Serious adverse events | 16 weeks
  Serious adverse events during the study period
Laboratory findings | 16 weeks
  Laboratory findings during the study period
Vital sign | 16 weeks
  Vital sign during the study period
Sirolimus blood concentration | Baseline, Week 4 and Week 12
  Blood concentration of Sirolimus is assessed by drug monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Mari Wataya-Kaneda, MD, PhD, Principal Investigator — Department of Dermatology, Graduate School of Medicine, Osaka University
Locations (1):
- Graduate School of Medicine, Osaka University, Suita, Osaka, Japan

REFERENCES:
- [Derived] Wataya-Kaneda M, Ohno Y, Fujita Y, Yokozeki H, Niizeki H, Ogai M, Fukai K, Nagai H, Yoshida Y, Hamada I, Hio T, Shimizu K, Murota H. Sirolimus Gel Treatment vs Placebo for Facial Angiofibromas in Patients With Tuberous Sclerosis Complex: A Randomized Clinical Trial. JAMA Dermatol. 2018 Jul 1;154(7):781-788. doi: 10.1001/jamadermatol.2018.1408. PMID 29800026